CLINICAL TRIAL: NCT02421172
Title: A Randomized, Double-blind, Placebo Controlled, Multiple Dose Study to Evaluate the Clinical Efficacy, Safety, Tolerability, Dose Relation, Pharmacokinetics and Pharmacodynamics of CJM112 in Moderate to Severe Chronic Hidradenitis Suppurativa Patients
Brief Title: Efficacy, Safety, and Pharmacokinetics Study of CJM112 in Hidradenitis Suppurativa Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCJM112X2202
Record Dates: First submitted 2015-03-18; First posted 2015-04-20 (Estimated); Results first posted 2019-05-23 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-06

CONDITIONS: Hidradenitis Suppurativa (Acne Inversa)
Keywords: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Period 1: CJM112 High Dose (Experimental): Period 1: CJM112 High Dose subcutaneously (s.c.) weekly for 5 doses followed by bi-weekly for 5 doses for a total of 10 doses
  Interventions: Biological: CJM112
- Period 1: Placebo (Placebo Comparator): Period 1: Placebo subcutaneously (s.c.) weekly for 5 doses followed by bi-weekly for 5 doses for a total of 10 doses
  Interventions: Drug: Placebo
- Period 2: CJM112 High Dose (Period 1) / Placebo (Period 2) (Placebo Comparator): Period 2: Placebo subcutaneously (s.c.) weekly for 5 doses then bi-weekly for 5 doses for a total of 10 doses this group.This group was on CJM112 High Dose in Period 1
  Interventions: Drug: Placebo
- Period 2: Placebo (Period 1)/CJM112 Low Dose (Period 2) (Experimental): Period 2: CJM112 Low Dose subcutaneously (s.c.) weekly for 5 doses then bi-weekly for 5 doses for a total of 10 doses this group.This group was on Placebo in Period 1
  Interventions: Biological: CJM112
- Period 2: Placebo (Period 1)/CJM112 High Dose (Period 2) (Experimental): Period 2: CJM112 High Dose subcutaneously (s.c.) weekly for 5 doses then bi-weekly for 5 doses for a total of 10 doses this group.This group was on Placebo in Period 1
  Interventions: Biological: CJM112

INTERVENTIONS:
Biological: CJM112 — CJM112 Fully human IgG1 monoclonal antibody
  Arms: Period 1: CJM112 High Dose; Period 2: Placebo (Period 1)/CJM112 High Dose (Period 2); Period 2: Placebo (Period 1)/CJM112 Low Dose (Period 2)
Drug: Placebo
  Arms: Period 1: Placebo; Period 2: CJM112 High Dose (Period 1) / Placebo (Period 2)

SUMMARY:
This is a randomized, double blind, multicenter study in patients with moderate to severe chronic hidradenitis suppurativa in parallel groups, to determine the efficacy and safety of multiple doses of CJM112 in comparison to placebo. The study has two periods to explore preliminary dose effects.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18 to 65 years of age with clinically diagnosed chronic HS for at least 1 year (prior to screening) who have undergone previous antibiotic therapy
2. Weight between 50 kg and 150 kg
3. HS-PGA score of at least moderate severity at the time of inclusion with at least 4 abscesses and/or nodules. HS lesions must be present in at least two distinct anatomical areas, and at least one area must be minimally Hurley Stage II (moderate)

Exclusion Criteria:

1. Use of previous biologics or other specified concomitant medications
2. Use of any systemic treatment for HS in the last 4 weeks prior to randomization
3. Presence of more than 25 draining fistulae.
4. Surgical treatment for HS in the last 4 weeks prior to randomization/first treatment.
5. Women of child-bearing potential and sexually active males unwilling to use a condom during intercourse while taking drug and for 15 weeks after stopping investigational medication.
6. Evidence of active tuberculosis at screening
7. History of severe systemic Candida infections or evidence of Candidiasis in the last two weeks
8. Active systemic or skin infections (other than common cold or HS related) during the two weeks before randomization/first treatment
9. Any live vaccines (including nasal spray flu vaccine) starting from 6 weeks before randomization.

Other protocol-defined inclusion/exclusion criteria may apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-04-13 (Actual); Primary Completion 2016-11-23 (Actual); Study Completion 2016-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R Hunger, Principal Investigator — University of Bern, Switzerland; Lars French, Principal Investigator — Zurich University Hospital, Switzerland; E P Prens, Principal Investigator — Erasmus MC, Rotterdam, Netherlands; Gregor Jemec, Principal Investigator — Dermatologisk Afdeling, Roskilde, Denmark; Sylke Schneider-Burrus, Principal Investigator — Psoriasis Research and Treatment Center, Charité hospital, Berlin, Germany; Christos C Zouboulis, Principal Investigator — Dessau Medical Center, Department of Dermatology, Venerology, Allergology and Immunology, Germany; Falk G Bechara, Principal Investigator — Ruhr-University Bochum, Germany; Barbara Horváth, Principal Investigator — University Medical Center Groningen, NL; Jan Mekkes, Principal Investigator — Dermatologie AMC, Amsterdam, NL; Christian Vestergaard, Principal Investigator — Dermato-verenologisk afdeling S, Denmark
Locations (16):
- United States (9):
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Ormond Beach, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Rockville, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Nashville, Tennessee
- Novartis Investigative Site, Roskilde, Denmark
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
- Netherlands (2):
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Rotterdam
- Switzerland (2):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Zurich

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study with 4 wks screening,two sequential treatment periods 16 wks (Period 1 & Extension Period 2)& 12 wks Follow-up. Randomization 2:1:1 to three sequences:Seq. 1: Period 1: CJM112 High Dose sc then Period 2: placebo sc; Seq. 2: Period 1: Placebo sc then Period 2: CJM112 Low Dose sc; Seq, 3: Period 1: Placebo sc then Period 2: CJM112 High Dose sc
Pre-assignment Details: A total of 66 patients were enrolled, randomized and entered into two sequential periods (Period 1 and Extension Period 2) of which 60 patients completed Week 16 in Period 1 and entered Extension Period 2.
Groups:
- Period 1: CJM112 High Dose: Period 1: CJM112 300mg subcutaneously (s.c.) weekly for 5 doses followed by bi-weekly for 5 doses for a total of 10 doses
- Extension Period 2: CJM112 High Dose /Placebo: Extension Period 2: Placebo subcutaneously (s.c.) weekly for 5 doses followed by bi-weekly for 5 doses for a total of 10 doses this group. This group was on CJM112 High Dose in Period 1
- Extension Period 2: Placebo/CJM112 Low Dose: Extension Period 2: CJM112 50mg subcutaneously (s.c.) weekly for 5 doses followed by bi-weekly for 5 doses for a total of 10 doses this group. This group was on Placebo in Period 1
- Extension Period 2: Placebo/CJM112 High Dose: Extension Period 2: CJM112 300mg subcutaneously (s.c.) weekly for 5 doses followed by bi-weekly for 5 doses for a total of 10 doses this group. This group was on Placebo in Period 1
Period: Period 1
Arm/Group | Period 1: CJM112 High Dose | Period 1: Placebo | Extension Period 2: CJM112 High Dose /Placebo | Extension Period 2: Placebo/CJM112 Low Dose | Extension Period 2: Placebo/CJM112 High Dose
Started | 33 | 33 | 0 | 0 | 0
PD Analysis Set Period 1 | 31 | 33 | 0 | 0 | 0
PK Analysis Set Period 1 | 33 | 0 | 0 | 0 | 0
Completed | 29 | 31 | 0 | 0 | 0
Not Completed | 4 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 1 | 0 | 0 | 0
Not completed — Patient/guardian decision | 0 | 1 | 0 | 0 | 0
Period: Period 2
Arm/Group | Period 1: CJM112 High Dose | Period 1: Placebo | Extension Period 2: CJM112 High Dose /Placebo | Extension Period 2: Placebo/CJM112 Low Dose | Extension Period 2: Placebo/CJM112 High Dose
Started | 0 | 0 | 29 | 16 | 15
Completed | 0 | 0 | 22 | 13 | 14
Not Completed | 0 | 0 | 7 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 4 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Patient/guardian decision | 0 | 0 | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Period 1: CJM112 High Dose | Period 1: Placebo | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (9.8) | 39 (10.9) | 37 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Clinical Responder Rate at Period 1: Week 16
Description: Proportion of study participants achieving a clinical response in Hidradenitis Suppurativa - Physician Global Assessment (HS-PGA) score An HS-PGA responder in period 1 was a participant who had an initial HS-PGA score of at least 3 at baseline (Day 1, inclusion criterion) that decreased by at least 2 points. The six-point Physician Global Assessment (PGA) (scores range from 0-5) based on the number of HS lesions ranges from clear to very severe.
Time Frame: Week 16
Population: PD analysis set 1 includes all patients who were CJM112-treated or placebo-treated in Period 1 with available PD data and no protocol deviations with relevant impact on PD data in Period 1.
Measure: Number; unit: participants
Arm/Group | Period 1: CJM112 High Dose | Period 1: Placebo
Number analyzed (Participants) | 31 | 32
participants | 10 | 4
Statistical Analysis 1: Comparison: Period 1: CJM112 High Dose vs Period 1: Placebo; Test type: Superiority or Other; Posterior probablility = 0.9729

2. Secondary Outcome: Clinical Responder Rate Period 1 at Week 2, 4, 8 and 12
Description: Proportion of study participants achieving a clinical response in Hidradenitis Suppurativa - Physician Global Assessment (HS-PGA) score A HS-PGA responder in Period 1 is a study participant who had an initial HS-PGA score of at least 3 at Baseline (Day 1, inclusion criterion) that decreased by at least 2 points. The six-point Physician Global Assessment (PGA) (scores range from 0-5) based on the number of HS lesions ranges from clear to very severe.
Time Frame: Week 2, 4, 8 and 12
Population: as for outcome 1
Measure: Number; unit: count of participants
Arm/Group | Period 1: CJM112 High Dose | Period 1: Placebo
Number analyzed (Participants) | 31 | 32
count of participants
  Week 2 | 4 | 3
  Week 4 | 6 | 3
  Week 8 | 5 | 6
  Week 12 | 7 | 4

3. Secondary Outcome: Pharmacokinetics (PK): Ctrough for CJM112 Period 1 and Period 2
Description: Ctrough is the serum concentration that is just prior to the beginning of, or at the end, of a dosing interval (mass/volume) for Period 1 (week 16) and Period 2/End of Study (week 44)
Time Frame: Week 16 and Week 44
Population: PK analysis set 1 includes all patients who were CJM112-treated in Period 1 with available PK data & no protocol deviations with relevant impact on PK data. PK analysis set 2 & 3 includes all patients from safety analysis set 2 & set 3 with available PK data & no protocol deviations with relevant impact on PK data for Period 2/End of Study.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Period 1: CJM112 High Dose | Extension Period 2: Placebo/CJM112 Low Dose | Extension Period 2: Placebo/CJM112 High Dose
Number analyzed (Participants) | 28 | 13 | 14
ug/mL | 21.4 (11.6) | 3.1 (2.6) | 24.4 (19.0)

4. Secondary Outcome: Pharmacokinetic Profile: T1/2 The Terminal Elimination Half-life for Period 1 & Period 2/End of Study
Description: T1/2 The terminal elimination half-life for Period 1 (Week 16) and Period 2/End of Study (Week 44)
Time Frame: Week 16 (period 1), Week 44 (End of Study Period 2)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Period 1: CJM112 High Dose | Extension Period 2: Placebo/CJM112 Low Dose | Extension Period 2: Placebo/CJM112 High Dose
Number analyzed (Participants) | 31 | 16 | 15
days | 16.09 (3.500) | 22.81 (0) | 19.85 (3.807)

5. Secondary Outcome: Immunogenicity - Incidence of ADA-positive and ADA-negative in Participants With or Without Pre-existing Antibodies in Period 1 and Period 2/End of Study
Description: Immunogenicity - Incidence of semi-quantitative determination of anti-CJM112 antibodies or ADAs. ADA-positive and ADA-negative in participants with or without pre-existing antibodies Period 1 (week 16) and Period 2/End of Study (week 44)
Time Frame: Week 16 (period 1), Week 44 (End of Study Period 2)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Period 1: CJM112 High Dose | Extension Period 2: Placebo/CJM112 Low Dose | Extension Period 2: Placebo/CJM112 High Dose
Number analyzed (Participants) | 33 | 16 | 15
participants
  Pre-existing Antibodies ADA negative | 2 | 1 | 7
  Pre-existing Antibodies ADA positive | 1 | 1 | 0
  NO Pre-existing Antibodies ADA negative | 21 | 10 | 9
  NO Pre-existing Antibodies ADA positive | 9 | 4 | 1

6. Secondary Outcome: Total Interleukin-17A (IL-17A Homodimer) in Serum at Pre-dose and Post-dose for Period 1 & Period 2
Description: Total Interleukin-17A (IL-17A homodimer) in serum at Pre-dose Period 1 (Day 1) & Pre-dose Period 2 (Day 113) and Post-dose Period 1 (Day 99) and Post-dose Period 2 (Day 211)
Time Frame: Pre-dose (Period 1 Day 1 & Period 2 Day 113), Post-dose Period 1(Day 99) and post-dose Period 2 (Day 211)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Period 1: CJM112 High Dose | Extension Period 2: Placebo/CJM112 Low Dose | Extension Period 2: Placebo/CJM112 High Dose
Number analyzed (Participants) | 33 | 16 | 15
pg/mL
  Pre-dose: number analyzed (Participants) | 32 | 16 | 14
  Pre-dose | 361 (2010) | 163 (647) | 158 (372)
  Post-dose: number analyzed (Participants) | 28 | 13 | 14
  Post-dose | 1160 (3190) | 943 (583) | 821 (538)

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All adverse events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit - End of Study Week 44.
Arm/Group | Period 1: CJM112 High Dose | Period 1: Placebo | Extension Period 2: CJM112 High Dose /Placebo | Extension Period 2: Placebo/CJM112 Low Dose | Extension Period 2: Placebo/CJM112 High Dose
Serious Adverse Events (participants affected / at risk) | 0/33 | 1/33 | 1/29 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 25/33 | 23/33 | 20/29 | 13/16 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: CJM112 High Dose (N=33) | Period 1: Placebo (N=33) | Extension Period 2: CJM112 High Dose /Placebo (N=29) | Extension Period 2: Placebo/CJM112 Low Dose (N=16) | Extension Period 2: Placebo/CJM112 High Dose (N=15)
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: CJM112 High Dose (N=33) | Period 1: Placebo (N=33) | Extension Period 2: CJM112 High Dose /Placebo (N=29) | Extension Period 2: Placebo/CJM112 Low Dose (N=16) | Extension Period 2: Placebo/CJM112 High Dose (N=15)
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eyelid cyst (Eye disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 5 | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 5 | 3 | 2 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 3 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0
Fatigue (General disorders) | 3 | 1 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 1 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 1 | 2 | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 1 | 3 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 1 | 0
Conjunctivitis (Infections and infestations) | 2 | 0 | 1 | 0 | 1
Cystitis (Infections and infestations) | 3 | 0 | 1 | 0 | 0
Eyelid infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 3 | 0 | 1 | 0
Influenza (Infections and infestations) | 3 | 1 | 2 | 0 | 1
Nasopharyngitis (Infections and infestations) | 7 | 4 | 4 | 2 | 3
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 1 | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 1 | 1 | 0
QRS axis abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
White blood cells urine (Investigations) | 0 | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 2 | 3 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 1 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 2
Intertrigo (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single- site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.